CLINICAL TRIAL: NCT03367260
Title: The Treatment Preferences of Women Diagnosed With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00080624
Record Dates: First submitted 2017-11-20; First posted 2017-12-08 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: patient preferences
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preference Elicitation — Survey of patient preferences for treatment

SUMMARY:
The primary objective of this study is to apply best-practice stated-preference methods to quantify the extent to which women with ovarian cancer accept the risks, side effects, and out-of-pocket costs associated with treatment in return for progression-free survival benefit afforded by a treatment, regardless of whether there is an overall survival benefit.

DETAILED DESCRIPTION:
The investigators propose to perform a preferences survey to be administered to women with ovarian cancer.The investigators anticipate that about 1/3 of the study cohort will include patients who are receiving treatment with an oral ADP-ribose polymerase inhibitors (PARPi). The investigators will begin by conducting interviews with 5 pilot subjects as they test the preferences survey. Based on their feedback the survey may be updated for clarity. During the final survey phase, subjects will be recruited and invited to participate in the choice experiment by Biologics, Inc., a specialty pharmacy company that dispenses oral PARPis. Subjects may also be recruited through ResearchMatch.org and at the Gynecologic Oncology division at Duke. Up to 300 women may be included in this study, at least 100 women will have received treatment with a PARPi.

Discrete choice experiment (DCE) questions generate limited dependent-variable, cross-section/time-series data. The study team will use random-parameters logit (RPL) to analyze the choice-format conjoint data collected in the DCE survey. Unobserved variation in preferences across the sample can bias estimates in conventional conditional-logit choice models. RPL avoids this potential bias by estimating a distribution of preferences around each model parameter that accounts for variations among individual preferences not accounted for by the variables in the model. The flexible correlation structure of RPL also accounts for within-sample correlation in the question sequence for each respondent.

There are no physical risks to subject participation in this survey protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian, fallopian tube, or primary peritoneal cancer

Exclusion Criteria:

* Does not read and understand English

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum on 300 subjects will be enrolled on this study. All subjects will have been diagnosed with ovarian, fallopian tube, or primary peritoneal cancer and at least 100 of them will have been treated with a PARPi.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Preference between two treatment alternatives as measured by discrete choice experiment (DCE). | baseline
  In the DCE, women are asked to choose between two hypothetical treatment scenarios characterized using 7 attributes (treatment schedule, out of pocket cost, peripheral neuropathy, nausea and vomiting, fatigue, progression-free survival and overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States